CLINICAL TRIAL: NCT06450964
Title: Establishment of Reproductive Cohort and Prediction Model of Genetic Counseling for Mitochondrial Genetic Diseases
Status: Enrolling by invitation | Type: Observational
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Dongmei Ji, Principal Investigator, Anhui Medical University
Other Study IDs: PJ2024-02-22
Record Dates: First submitted 2024-06-03; First posted 2024-06-10 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-06

CONDITIONS: Mitochondrial Diseases
Keywords: mitochondrial diseases; mitochondrial DNA mutation; reproductive cohort; genetic counseling
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, oral epithelial cells, fingernail, trophectoderm cells, embryo culture medium, amniotic fluid, placenta, granulosa cell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Biological samples such as blood, urine, oral epithelial cells and nails of carriers were collected, and the mitochondrial DNA mutation heterogeneity level was determined. — Biological samples such as blood, urine, oral epithelial cells and nails of carriers were collected, and some granulosa cells, trophoderm cells, embryo culture fluid, embryo biopsy fluid, and embryo trophoblast cells were collected. Placenta and umbilical cord blood samples of some fetuses were collected after delivery, and the mitochondrial DNA mutation heterogeneity level was determined.

SUMMARY:
The goal of this observational study is to provide a reference for clinicians to conduct genetic counseling and carry out preimplantation genetic testing of mitochondrial patients. The main questions it aims to answer are:

* The relationship between mitochondrial mutation load and clinical symptom
* The symptomatic threshold of common mitochondrial DNA mutations
* The distribution of mitochondrial mutation load in offspring and genetic rule of mitochondrial DNA mutation
* The minimum number of eggs taken by preimplantation genetic testing in mitochondrial mutation carriers Biological samples such as blood, urine, oral epithelial cells, nails, some granulosa cells, trophoderm cells, embryo culture fluid, embryo biopsy fluid, and embryo trophoblast cells of the participants will be collected and the mutation loads of them will be measured. The clinical symptoms and mutation load of the participants will be followed up once a year.

DETAILED DESCRIPTION:
A total of 600 carriers of disease-causing mitochondrial DNA mutations will be selected as the research objects. The basic information, reproductive history, clinical and genetic diagnosis, and clinical symptoms of the carriers will be investigated by questionnaire. Biological samples such as blood, urine, oral epithelial cells, nails, some granulosa cells, trophoderm cells, embryo culture fluid, embryo biopsy fluid, and embryo trophoblast cells of the participants will be collected and the mutation loads of them will be measured. Placenta and umbilical cord blood samples of some fetuses will be collected after delivery, and the mitochondrial DNA mutation heterogeneity level will be determined. Multiple Logistic regression, Sewell-Wright equation, Kimura equation, binomial distribution model, and machine learning model will be used to establish a prediction model of the incidence probability of mitochondrial diseases and predict the onset threshold of common mitochondrial DNA mutations after standardizing. The distribution model of mitochondrial mutation load in offspring will be established to predict the maternal genetic risk of mitochondrial DNA mutation. A prediction model for egg retrieval will be established to estimate the minimum number of eggs taken by preimplantation genetic testing in mitochondrial mutation carriers. Finally, an online prediction platform for mitochondrial genetic disease genetic counseling will be established to provide standardized standards for mitochondrial disease genetic counseling and PGT.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mitochondrial DNA diseases

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: mtDNA mutation carriers from The First Affiliated Hospital of Anhui Medical University
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms of mitochondrial disease | 3 years
  The enrolled patients were followed up once a year. Symptoms that the patient has due to mitochondrial DNA mutations are recorded.

SECONDARY OUTCOMES:
level of mitochondrial DNA mutation | 3 years
  The enrolled patients were followed up once a year. Levels of mitochondrial DNA mutation are measured by next generation sequencing and ddPCR.
Tissue-specific distribution of mitochondrial DNA mutation levels | When they enrolled
  The levels of mitochondrial DNA mutations in blood, urine, oral epithelial cells, nails, etc. were measured when the patients were enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, Dr., Study Chair — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided